CLINICAL TRIAL: NCT03386071
Title: Individual Patient Program for Patient With Progressive Metastatic Castrate Resistant Prostate Cancer; Monotherapy Treatment With Trametinib
Brief Title: Compassionate Use: Progressive Metastatic Castrate Resistant Prostate Cancer; Monotherapy Treatment With Trametinib
Status: No longer available | Type: Expanded Access
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: 17-001886; Compassionate Use Trametinib (Other: Jonsson Comprehensieve Cancer Center)
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Progressive Metastatic Castrate Resistant Prostate Cancer
MeSH Terms: interventions — trametinib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Trametinib 2 mg — The dosage of trametinib for oral administration is 2mg once daily.

SUMMARY:
The dosage of trametinib for oral administration is 2mg once daily. The patient is instructed to take the trametinib oncedaily dose at approximately the same time each day, by mouth with approximately 200 mL (almost 1 cup) of water on an empty stomach, either 1 hour before or 2 hours after a meal.

DETAILED DESCRIPTION:
The dosage of trametinib for oral administration is 2mg once daily. The patient is instructed to take the trametinib once daily dose at approximately the same time each day, by mouth with approximately 200 mL (almost 1 cup) of water on an empty stomach, either 1 hour before or 2 hours after a meal.

The patient will be provided with complete dosing instructions from his treating physician. If the subject is instructed that if he vomits after taking either of the medications provided under this program, he should not retake the dose. The patient should take the next dose as originally scheduled. If a dose is missed, the patient should not double the next regularly scheduled dose. However, the patient can take the missed dose immediately if the next scheduled dose is at least 12 hours later. If the next scheduled dose is due in less than 12 hours, the patient is instructed to skip the dose and resume dosing the next day at the regular time. Then to take the next dose at the usual time the subject is scheduled to take it. It is not known for how long the subject will remain in the program because each patient may respond differently to the treatment. The length of time the patient will take trametinib therapy will depend on his cancer status and how well he tolerates the drugs. If he experiences severe side effects, he is instructed to call his treating physician immediately. The treating physician may advise him stop compassionate used of trametinib or may advise him to lower the dose. Trametinib may also be stopped completely at his Treating Physician's discretion. The treating physician will use his/her clinical expertise considering the intensity of the adverse effect and/or the results of your laboratory tests to make his/her decision. The Treating Physician may consult with the Novartis Country Pharma Organization Medical Advisor/Director about dose interruptions or modifications.

ELIGIBILITY:
Inclusion Criteria:

* Progressive Metastatic Castrate Resistant Prostate Cancer

Exclusion Criteria:

* Absence of Progressive Metastatic Castrate Resistant Prostate Cancer

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Rettig, M.D., Principal Investigator — Jonsson Comprehensieve Cancer Center